CLINICAL TRIAL: NCT02670837
Title: Study of Epidermal Grafting Using the CelluTome Epidermal Harvesting System for the Treatment of Individual Lesions in Persons With Epidermolysis Bullosa [MT2015-36]
Brief Title: Study of Cellutome System for Treatment of Individual Lesions in EB Pts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015LS154
Record Dates: First submitted 2016-01-08; First posted 2016-02-02 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Graft from HCT donor (Experimental): Cells are harvested from a donor using Cellutome, then transferred via Adaptic dressing to the recipient's wound with up to 3 donor harvest sites/treated wound sites on day 0.
  Interventions: Device: Cellutome Epidermal Harvesting System
- Self donor from intact skin patch (Experimental): Cells are harvested from the subject using Cellutome, then transferred via Adaptic dressing to that subject's wound with up to 3 harvest sites/treated wound sites on day 0.
  Interventions: Device: Cellutome Epidermal Harvesting System

INTERVENTIONS:
Device: Cellutome Epidermal Harvesting System

SUMMARY:
Few but persistent wounds often remain even after successful hematopoietic cell transplantation for systemic genodermatosis epidermolysis bullosa (EB). The investigators propose local wound therapy using epidermal skin grafting from the same donor that provided the hematopoietic graft, or from the same EB individual with a mosaic (naturally gene corrected) skin. In both cases permissive immune system and skin chimerism is expected to enable long-term epidermal engraftment and wound healing. The investigators will use FDA approved vacuum device (CelluTome®, Regulation number 878.4820) that enables scar-free harvesting of epidermis and its transfer on a non-adherent silicone dressing (Adaptic) to the recipient as a wound dressing.

ELIGIBILITY:
Inclusion Criteria:

Patient (Recipient)

* Diagnosis of Dystrophic Epidermolysis Bullosa (DEB) or Junctional Epidermolysis Bullosa (JEB) with at least one wound, visibly free from infection (or previously treated) and meets the eligibility for Arm A or Arm B based on the skin graft source:
* Cell harvest from previous hematopoietic cell transplantation (HCT) donor (Arm A) - not applicable if Arm B

  * At least 6 months after hematopoietic cell transplantation with donor chimerism

    * Peripheral blood donor chimerism should be measured within 21 days of grafting and be >/= 5% and stable. Stability of chimerism will be determined by the protocol team and based on 3 peripheral blood chimerism values at least 1 month apart.
  * No history of pre-BMT autoimmune cytopenias
  * Off immune suppressive therapy
  * Original transplant donor is available and willing to be the epidermis donor
* Self-donation (Arm B) - not applicable if Arm A

  * Proven somatic reversion
  * Site for skin grafting free of cellulitis and any other clinically evident abnormalities
  * Meets donor eligibility
* Insurance pre-authorization for procedure, if applicable
* Voluntary written consent (patient or parent/guardian for minors with assent) prior to any research related procedures or treatment.

Skin Graft Donor (either hematopoietic cell transplantation donor for the EB patient [Arm A] or EB patient herself/himself [Arm B])

* Age > 2 years (based on prior safety testing of the device)
* Healthy on physical examination in the opinion of the evaluating provider
* Negativity for Hepatitis B and C, HIV, and HTLV1/2 within 30 days of donation
* Voluntary written consent (donor or parent/guardian for minors with assent) prior to any research related procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christen Ebens, MD, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center and Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Ebens CL, McGrath JA, Riedl JA, Keith AR, Lilja G, Rusch S, Keene DR, Tufa SF, Riddle MJ, Shanley R, Van Heest AE, Tolar J. Immune tolerance of allogeneic haematopoietic cell transplantation supports donor epidermal grafting of recessive dystrophic epidermolysis bullosa chronic wounds. Br J Dermatol. 2021 Jun;184(6):1161-1169. doi: 10.1111/bjd.19503. Epub 2020 Dec 14. PMID 32866988

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: grafts
Groups:
- Graft From HCT Donor; Self-Donor: Cells are harvested from a donor using Cellutome, then transferred via Adaptic dressing to the recipient's wound with up to 3 donor harvest sites/treated wound sites on day 0.
  Cellutome Epidermal Harvesting System
- Donor: Cells are harvested from a donor using Cellutome, then transferred via Adaptic dressing to the recipient's wound.
  Cellutome Epidermal Harvesting System
Period: Overall Study
Arm/Group | Graft From HCT Donor | Donor | Self-Donor
Started | 17; 51 grafts | 17; 0 grafts | 0; 0 grafts (3 participants screened for self-donor arm were not eligible.)
Completed | 15; 45 grafts | 17; 0 grafts | 0; 0 grafts
Not Completed | 2; 6 grafts | 0; 0 grafts | 0; 0 grafts
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donor: Cells are harvested from a donor using Cellutome, then transferred via Adaptic dressing to the recipient's wound with up to 3 donor harvest sites/treated wound sites on day 0.
  Cellutome Epidermal Harvesting System
- Total: Total of all reporting groups
Arm/Group | Graft From HCT Donor | Donor | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 10 | 25
  Between 18 and 65 years | 2 | 7 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Grafts Successfully Treated
Description: If the body surface area affected by the wound is at least 50%
  lower at 12 weeks relative to baseline, the graft will be considered
  successful.
Time Frame: 12 weeks after grafting
Measure: Number (95% Confidence Interval); unit: Percentage of grafts
Units Other Than Participants: grafts
Arm/Group | Graft From HCT Donor
Number analyzed (Participants) | 15
Number analyzed (grafts) | 45
Percentage of grafts | 78 [63 to 89]

2. Secondary Outcome: Participants With Lesion Free Skin
Description: Participants without Squamous cell carcinoma (SCC) at graft site. Wound reassessments will be performed via photographs and follow-up visits.
Time Frame: 1 year after grafting
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Graft From HCT Donor
Number analyzed (Participants) | 15
Percentage of participants | 100 [80 to 100]

3. Secondary Outcome: Longevity of Grafted Skin
Description: Percentage of patients who have had a 6 week period of lesion free skin by the time they are 1 year post grafting. Wound reassessments will be performed via photographs and follow-up visits.
Time Frame: 1 year after grafting
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Graft From HCT Donor
Number analyzed (Participants) | 15
Percentage of participants | 34 [21 to 50]

4. Secondary Outcome: Percentage Change of a Patient's IScorEB Assessment Score
Description: Measure percent of changes in quality of life (QOL) through pain, itching, and general QOL IScorEB questionnaire. Scores can range from 16 to 112. The QOLS scores are summed so that a higher score indicates higher quality of life.
Time Frame: Baseline and 6 weeks
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Graft From HCT Donor
Number analyzed (Participants) | 13
Percent change
  Change in pain QOL score | -2.1 [-31.5 to 27.3]
  Change in itch QOL score | -1.9 [-33.9 to 30.1]
  Change in General QOL score | 3.1 [-13.7 to 19.8]

5. Secondary Outcome: Percentage Change of a Patient's IScoreEB Assessment Score
Description: as for outcome 4
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Graft From HCT Donor
Number analyzed (Participants) | 12
Percent change
  Change in pain QOL score | -8.1 [-32.5 to 16.3]
  Change in itch QOL score | -10.4 [-50.1 to 29.2]
  Change in general QOL score | -0.4 [-18 to 17.2]

6. Secondary Outcome: Scar-free Healing of the Body Sites of the Donor
Description: Percentage of donors with no evidence of non-healed skin. Wound reassessments will be performed via photographs and follow-up visits.
Time Frame: 1 year after grafting
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Donor
Number analyzed (Participants) | 17
Percentage of participants | 100 [80 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Donor: Cells are harvested from a donor using Cellutome, then transferred via Adaptic dressing to the recipient's wound.
Arm/Group | Graft From HCT Donor | Donor
All-Cause Mortality (participants affected / at risk) | 2/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT02670837/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT02670837/ICF_001.pdf